CLINICAL TRIAL: NCT07383896
Title: Chronic Obstructive Pulmonary Disease and Asthma in Workers at Navanakorn Industrial Zone, Thailand
Status: Recruiting | Type: Observational
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Other Study IDs: MTU-EC-IM-1-024/68
Record Dates: First submitted 2026-01-18; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Asthma; COPD
Keywords: asthma; COPD; pulmonary function; worker; industry; Thailand
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Workers: Workers aged 18 years or older at Navanakorn industrial zone, Thailand
  Interventions: Diagnostic Test: Pulmonary function test

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — Spirometry with bronchondilator test will be performed.

SUMMARY:
The goal of this observational study is to determine the prevalence of asthma and chronic obstructive pulmonary disease (COPD) among workers in an industrial zone in Thailand.

The main question the study aims to answer is:

What is the prevalence of asthma and COPD among workers in Thailand? Participants will complete a questionnaire on respiratory symptoms and undergo pulmonary function testing.

DETAILED DESCRIPTION:
This study is a cross-sectional study. The study aims to determine the prevalence of asthma and COPD among workers in the Navanakorn Industrial Zone, Thailand. Thai subjects aged 18 years or older are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older

Exclusion Criteria:

* Inability to perform spirometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18 years or older who work or live in the Navanakorn Industrial Zone, Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of asthma among workers at the Navanakorn Industrial Zone | Baseline
  Prevalence rate of asthma among workers in the Navanakorn Industrial Zone
Prevalence of COPD among workers in the Navanakorn Industrial Zone | Baseline
  Prevalence rate of COPD among workers in the Navanakorn Industrial Zone

SECONDARY OUTCOMES:
Prevalence of abnormal lung function among workers in the Navanakorn Industrial Zone | Baseline
  Prevalence rate of abnormal lung function among workers in the Navanakorn Industrial Zone

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Faculty of Medicine, Thammasat University, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and documents will be available for sharing immediately after publication for a period of 2 years.

REFERENCES:
- [Result] Vested A, Kolstad HA, Basinas I, Burdorf A, Elholm G, Heederik D, Jacobsen GH, Kromhout H, Omland O, Schaumburg I, Sigsgaard T, Vestergaard JM, Wouters IM, Schlunssen V. Dust exposure and the impact on hospital readmission of farming and wood industry workers for asthma and chronic obstructive pulmonary disease (COPD). Scand J Work Environ Health. 2021 Mar 1;47(2):163-168. doi: 10.5271/sjweh.3926. Epub 2020 Oct 19. PMID 33073852
- [Result] Garg R, Matreja PS, Maqusood M. Analysis of lung function and respiratory symptoms in brass/metal industrial workers of Moradabad, Uttar Pradesh, India. Ann Afr Med. 2023 Apr-Jun;22(2):219-223. doi: 10.4103/aam.aam_24_22. PMID 37026203
- [Result] Bansal N, Lanjewar A, Acharya S, Shukla S. Assessment of pulmonary function test in brick factory workers. J Family Med Prim Care. 2022 Nov;11(11):6916-6919. doi: 10.4103/jfmpc.jfmpc_504_22. Epub 2022 Dec 16. PMID 36993005
- [Result] Rafeemanesh E, Alizadeh A, Afshari Saleh L, Zakeri H. A study on respiratory problems and pulmonary function indexes among cement industry workers in Mashhad, Iran. Med Pr. 2015;66(4):471-7. doi: 10.13075/mp.5893.00115. PMID 26536964
- [Result] Nasri SM, Putri FA, Sunarno S, Fauzia S, Ramdhan DH. PM2.5 exposure and lung function impairment among fiber-cement industry workers. J Public Health Res. 2023 Jan 13;12(1):22799036221148989. doi: 10.1177/22799036221148989. eCollection 2023 Jan. PMID 36654813
- [Result] Elshaer N, Foda N, Shehata S. Respiratory symptoms and pulmonary function impairment among textile industry workers in Alexandria, Egypt. J Public Health Afr. 2023 Oct 1;14(10):2741. doi: 10.4081/jphia.2023.2741. eCollection 2023 Oct 31. PMID 38020280
- [Result] Papageorgiou CV, Savourdos P, Douna E, Georgakopoulou VE, Makrodimitri S, Dounias G. Respiratory Symptoms and Pulmonary Function of Workers in the Waste Management Industry. Cureus. 2021 Aug 9;13(8):e17027. doi: 10.7759/cureus.17027. eCollection 2021 Aug. PMID 34522508
- [Result] Cox-Ganser JM, White SK, Fedan KB, Bailey RL, Fechter-Leggett E, Cummings KJ. Spirometric Abnormalities and Lung Function Decline in Current and Former Microwave Popcorn and Current Flavoring Manufacturing Workers. J Occup Environ Med. 2020 Jun;62(6):412-419. doi: 10.1097/JOM.0000000000001860. PMID 32510907
- [Result] Boonsawat W, Charoenphan P, Kiatboonsri S, Wongtim S, Viriyachaiyo V, Pothirat C, Thanomsieng N. Survey of asthma control in Thailand. Respirology. 2004 Aug;9(3):373-8. doi: 10.1111/j.1440-1843.2004.00584.x. PMID 15363011
- [Result] Saiphoklang N, Ruchiwit P, Kanitsap A, Tantiyavarong P, Vatcharavongvan P, Palungrit S, Leelasittikul K, Pugongchai A, Poachanukoon O. Prevalence of Chronic Obstructive Pulmonary Disease and Asthma in the Community of Pathumthani, Thailand. Diseases. 2025 Apr 23;13(5):130. doi: 10.3390/diseases13050130. PMID 40422562
- [Result] Saiphoklang N, Ruchiwit P, Kanitsap A, Tantiyavarong P, Vatcharavongvan P, Palungrit S, Leelasittikul K, Pugongchai A, Poachanukoon O. Silicosis and Pulmonary Functions Among Residents Exposed to Dust in Saraburi Thailand. Diseases. 2025 Nov 13;13(11):372. doi: 10.3390/diseases13110372. PMID 41294912